CLINICAL TRIAL: NCT05082324
Title: Evaluation of Modification in VO2 Max After Performing the PAPS 53 Program
Brief Title: Evaluation of Modification in VO2 Max After Performing the "Physical Activity and Health Course (PAPS) 53" Program
Acronym: EVOP-53
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 49RC21_0332
Record Dates: First submitted 2021-10-01; First posted 2021-10-18 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Cardio-Respiratory Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adapted physical activity (Experimental)
  Interventions: Other: Adapted physical activity

INTERVENTIONS:
Other: Adapted physical activity — Patient participates in an adapted physical activity program for 3 months, with 2 one-hour sports sessions per week

SUMMARY:
Physical inactivity is the leading cause of preventable death in developed countries, ahead of smoking. It is responsible for 5.3 million (9%) of the 57 million deaths worldwide in 2008 and 10% of deaths in Europe.

Encouraging regular physical activity in the general population is a public health priority.

Cardiorespiratory capacity, measured during an exercise test, expressed as maximal oxygen consumption (VO2 max) or Metabolic Equivalent Task (MET) = oxygen consumption at rest [3.5 ml/kg/min], is an excellent indicator of individual exercise capacity and is increased by regular physical activity (PA).

Any gain in cardiorespiratory capacity of 1 MET is accompanied by a 12% reduction in mortality whether the subjects are free of any cardiovascular pathology or have a chronic pathology, regardless of their age.

As physical activity is an integral part of the management of many diseases, it seems essential to evaluate specific protocols oriented towards the maintenance or development of strength or endurance, or even mixed protocols.

The PAPS 53 (Physical Activity and Health Pathway), set up in Mayenne, responds to the demand for prescription of adapted physical activity. It is a 3-month program with 2 one-hour sports sessions per week (30 minutes of endurance and 30 minutes of muscle strengthening).

The National Sport and Health Strategy 2019-2024 expert group recommends better defining the characteristics of physical activity (intensity, frequency, etc.) to determine the effect (dose-response) on different at-risk populations and according to the type of pathology.

Investigators proposed to study by comparison the VO2 max values obtained during the two exercise tests (at inclusion and after 3 months of physical activity program). The hypothesis is that, after completion of the PAPS program, the VO2 max value of a patient will be significantly increased.

The control group is represented by the patients who have not yet followed the adapted physical activity program. The intervention group is therefore composed of the same patients. The aim is to compare the same group of eligible patients, before and after having followed the "PAPS 53" protocol

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years)
* Patient integrating the PAPS 53 with an indication to perform a stress test
* Person affiliated or benefiting from a social security plan
* Patient having signed an informed consent beforehand

Exclusion Criteria:

* Contraindication to the performance of the stress test
* Patient unable to understand the objectives or instructions of the study
* Poor understanding of the French language
* Pregnant, nursing or parturient woman
* Person deprived of liberty by judicial or administrative decision
* Person under forced psychiatric care
* Person admitted to a health or social institution for purposes other than research research
* Person subject to a legal protection measure
* Person unable to express his or her consent
* Person in a period of exclusion relative to another intervention research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-04 (Estimated); Primary Completion 2022-05-04 (Estimated); Study Completion 2022-05-04 (Estimated)

PRIMARY OUTCOMES:
To assess maximal oxygen consumption (VO2 max) measured during an effort test | 3 month
  Effort test

SECONDARY OUTCOMES:
To assess the quality of life | 3 month
  Short Form-36; min value 36 and max value 149

CONTACTS AND LOCATIONS:
Locations (1):
- CH Laval, Laval, France